CLINICAL TRIAL: NCT04636801
Title: A 52-week, Randomized, Double-blind, Placebo-controlled, Parallel-group, Study to Evaluate the Efficacy and Safety of Two Doses of CHF6001 DPI add-on to Maintenance Triple Therapy in Subjects With Chronic Obstructive Pulmonary Disease (COPD) and Chronic Bronchitis
Brief Title: A 52-week, Placebo-controlled Study to Evaluate the Efficacy and Safety of 2 Doses of CHF6001 DPI (Tanimilast), as add-on to Maintenance Triple Therapy in Subjects With COPD and Chronic Bronchitis (PILASTER)
Acronym: PILASTER
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Strategic decision by Sponsor; not due to safety reasons
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLI-06001AA1-04; 2020-003666-40 (EudraCT Number)
Record Dates: First submitted 2020-11-16; First posted 2020-11-19 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Chronic Bronchitis; PDE4 inhibitor; anti-inflammatory respiratory drug; Tanimilast
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CHF6001 1600µg (Experimental)
  Interventions: Drug: Experimental: CHF6001 1600µg
- CHF6001 3200µg (Experimental)
  Interventions: Drug: Experimental: CHF6001 3200µg
- CHF6001 Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Experimental: CHF6001 1600µg — CHF6001 400µg, 2 inhalations bid (total daily dose of 1600µg).
  Arms: CHF6001 1600µg
Drug: Experimental: CHF6001 3200µg — CHF6001 800µg, 2 inhalations bid (total daily dose of 3200µg).
  Arms: CHF6001 3200µg
Drug: Placebo — CHF6001 matching placebo, 2 inhalations bid.
  Arms: CHF6001 Placebo

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of two doses of CHF6001 (Tanimilast), as add-on to maintenance triple therapy in the target patient population.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥ 40 years with COPD and chronic bronchitis
* Current or ex-smokers (history ≥ 10 pack years).
* Post-bronchodilator FEV1 <60% of the subject predicted normal value and FEV1/FVC ratio < 0.7.
* At least, one moderate or severe COPD exacerbation in previous year.
* CAT score ≥ 10
* Subjects on regular maintenance triple therapy for at least 12 months prior to screening and receiving regular maintenance triple therapy for at least 3 months prior to screening visit

Exclusion Criteria:

* Subjects with current asthma.
* Subjects with moderate or severe COPD exacerbation 4 weeks prior to study entry and randomization.
* Subjects with known α-1 antitrypsin deficiency as the underlying cause of COPD.
* Subjects with COPD emphysema or mixed phenotypes.
* Subjects with known respiratory disorders other than COPD.
* Subjects with active cancer or a history of lung cancer with full recovery less than 1 year after completing cancer therapy.
* Subjects under Roflumilast treatment within 6 months before study entry.
* Subjects with a diagnosis of depression, generalised anxiety disorder, suicidal ideation.
* Subjects with clinically significant cardiovascular.
* Subjects with a significant neurological disease.
* Subjects with clinically significant laboratory abnormalities.
* Subjects with moderate or severe hepatic impairment

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4710 (Actual)
Dates: Start 2021-07-14 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
The number of moderate and severe COPD exacerbations occurring during the planned 52-week treatment period. | Up to 52 weeks
  Moderate or severe exacerbation is defined by symptomatic worsening of COPD:
  * Moderate: requiring use of systemic corticosteroid (oral/IV/IM corticosteroids), and/or use of antibiotics
  * Severe: requiring hospitalisation or resulting in death

SECONDARY OUTCOMES:
The time to first moderate or severe exacerbation. | Up to 52 weeks
The annual rate of severe exacerbation. | Up to 52 weeks
The time to first severe exacerbation. | Up to 52 weeks
The number of on-treatment severe exacerbations. | Up to 52 weeks
Change from baseline (pre-dose visit 2) in pre-dose FEV1 at week 52. | At Week 52
Change from baseline in SGRQ total and domain scores at week 52. | At week 52
SGRQ response (change from baseline SGRQ total score ≤ -4) at week 52. | At week 52
Change from baseline to last inter-visit period (week 40-52) in E-RS Total and subscale scores | Up to 52 weeks
E-RS response (change from baseline E-RS Total score ≤ -2) at week 52. | At week 52
Change from baseline to last inter-visit period (week 40-52) in the percentage of days without intake of rescue medication and in the average rescue medication use (number of puffs) | Up to 52 weeks
Time to study medication discontinuation for any reason. | Up to 52 weeks
Time to moderate or severe exacerbation or study medication discontinuation due to any adverse event, lack of efficacy or death (composite endpoint) and time to study medication discontinuation component. | Up to 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Klaus F. Rabe, Prof., Principal Investigator — LungenClinic Grosshansdorf GmbH Wöhrendamm 80 22927 Großhansdorf GERMANY
Locations (447):
- United States (15):
  - Chiesi Clinical Trial - Site 840402, Sheffield, Alabama
  - Chiesi Clinical Trial - Site 840480, Northridge, California
  - Chiesi Clinical Trial - Site 840487, Cutler Bay, Florida
  - Chiesi Clinical Trial - Site 840404, Hollywood, Florida
  - Chiesi Clinical Trial - Site 840407, Miami, Florida
  - Chiesi Clinical Trial - Site 840444, Miami, Florida
  - Chiesi Clinical Trial - Site 840437, Miami, Florida
  - Chiesi Clinical Trial - Site 840403, Miami, Florida
  - Chiesi Clinical Trial - Site 840463, Orlando, Florida
  - Chiesi Clinical Trial - Site 840401, Peachtree Corners, Georgia
  - Chiesi Clinical Trial - Site 840478, New Windsor, New York
  - Chiesi Clinical Trial - Site 840483, Philadelphia, Pennsylvania
  - Chiesi Clinical Trial - Site 840474, Kerrville, Texas
  - Chiesi Clinical Trial - Site 840409, Plano, Texas
  - Chiesi Clinical Trial - Site 840481, San Antonio, Texas
- Albania (10):
  - Chiesi Clinical Trial - Site 8455, Durrës
  - Chiesi Clinical Trial - Site 8459, Durrës
  - Chiesi Clinical Trial - Site 8457, Elbasan
  - Chiesi Clinical Trial - Site 8460, Korçë
  - Chiesi Clinical Trial - Site 8451, Tirana
  - Chiesi Clinical Trial - Site 8452, Tirana
  - Chiesi Clinical Trial - Site 8453, Tirana
  - Chiesi Clinical Trial - Site 8454, Tirana
  - Chiesi Clinical Trial - Site 8456, Tirana
  - Chiesi Clinical Trial - Site 8458, Tirana
- Argentina (28):
  - Chiesi Clinical Trial - Site 32415, Buenos Aires
  - Chiesi Clinical Trial - Site 32407, Buenos Aires
  - Chiesi Clinical Trial - Site 32410, Buenos Aires
  - Chiesi Clinical Trial - Site 32454, Buenos Aires
  - Chiesi Clinical Trial - Site 32457, Caba
  - Chiesi Clinical Trial - Site 32459, CABA
  - Chiesi Clinical Trial - Site 32414, Ciudad Autonoma de Buenos Aire
  - Chiesi Clinical Trial - Site 32403, Córdoba
  - Chiesi Clinical Trial - Site 32409, Córdoba
  - Chiesi Clinical Trial - Site 32401, Florida
  - Centro de Medicina Respiratoria - Concepcion del Uruguay - site 32463, Forestal Entre Ríos
  - Chiesi Clinical Trial - Site 32455, La Plata
  - Chiesi Clinical Trial - Site 32458, Mar del Plata
  - Chiesi Clinical Trial - Site 32462, Mar del Plata
  - Chiesi Clinical Trial - Site 32405, Mendoza
  - Chiesi Clinical Trial - Site 32411, Mendoza
  - Chiesi Clinical Trial - Site 32413, Mendoza
  - Chiesi Clinical Trial - Site 32402, Monte Grande
  - Chiesi Clinical Trial - Site 32406, Quilmes
  - Chiesi Clinical Trial - Site 32453, Rosario
  - Chiesi Clinical Trial - Site 32460, San Fernando
  - Chiesi Clinical Trial - Site 32408, San Juan Bautista
  - Chiesi Clinical Trial - Site 32412, San Miguel de Tucumán
  - Chiesi Clinical Trial - Site 32451, San Miguel de Tucumán
  - Chiesi Clinical Trial - Site 32452, San Miguel de Tucumán
  - Chiesi Clinical Trial - Site 32461, San Miguel de Tucumán
  - Chiesi Clinical Trial - Site 32464, San Miguel de Tucumán
  - Chiesi Clinical Trial - Site 32456, Santa Fe
- Australia (6):
  - Chiesi Clinical Trial - Site 36453, Adelaide
  - Chiesi Clinical Trial - Site 36454, Box Hill
  - Chiesi Clinical Trial - Site 36455, Campbelltown
  - Chiesi Clinical Trial - Site 36456, Clayton
  - Chiesi Clinical Trial - Site 36451, South Brisbane
  - Chiesi Clinical Trial - Site 36452, Westmead
- Austria (6):
  - Chiesi Clinical Trial - Site 40402, Feldbach
  - Chiesi Clinical Trial - Site 40404, Grieskirchen
  - Chiesi Clinical Trial - Site 40406, Linz
  - Chiesi Clinical Trial - Site 40401, Linz
  - Chiesi Clinical Trial - Site 40403, Linz
  - Chiesi Clinical Trial - Site 40405, Wels
- Bosnia and Herzegovina (10):
  - Chiesi Clinical Trial - Site 070401, Banja Luka
  - Chiesi Clinical Trial - Site 070407, Doboj
  - Chiesi Clinical Trial - Site 070460, Mostar
  - Chiesi Clinical Trial - Site 070404, Pale
  - OJ Dom zdravlja Novo Sarajevo "Omer Maslić" - Site 70408, Sarajevo
  - Chiesi Clinical Trial - Site 070405, Sarajevo
  - Chiesi Clinical Trial - Site 070406, Sarajevo
  - Chiesi Clinical Trial - Site 070403, Tešanj
  - Chiesi Clinical Trial - Site 070402, Tuzla
  - Chiesi Clinical Trial - Site 070463, Tuzla
- Bulgaria (29):
  - Chiesi Clinical Trial - Site 100435, Blagoevgrad
  - Chiesi Clinical Trial - Site 100434, Dimitrovgrad
  - Chiesi Clinical Trial - Site 100453, Gabrovo
  - Chiesi Clinical Trial - Site 100423, Haskovo
  - Chiesi Clinical Trial - Site 100433, Kozloduy
  - Chiesi Clinical Trial - Site 100455, Lovech
  - Chiesi Clinical Trial - Site 100415, Montana
  - Chiesi Clinical Trial - Site 100432, Pernik
  - Chiesi Clinical Trial - Site 100422, Pleven
  - Chiesi Clinical Trial - Site 100452, Plovdiv
  - Chiesi Clinical Trial - Site 100456, Plovdiv
  - Chiesi Clinical Trial - Site 100437, Razgrad
  - Chiesi Clinical Trial - Site 100412, Rousse
  - Chiesi Clinical Trial - Site 100416, Rousse
  - Chiesi Clinical Trial - Site 100436, Sevlievo
  - Chiesi Clinical Trial - Site 100460, Sliven
  - Chiesi Clinical Trial - Site 100409, Sofia
  - Chiesi Clinical Trial - Site 100414, Sofia
  - Chiesi Clinical Trial - Site 100417, Sofia
  - Chiesi Clinical Trial - Site 100418, Sofia
  - Chiesi Clinical Trial - Site 100420, Sofia
  - Chiesi Clinical Trial - Site 100430, Sofia
  - Chiesi Clinical Trial - Site 100431, Sofia
  - Chiesi Clinical Trial - Site 100438, Sofia
  - Chiesi Clinical Trial - Site 100424, Stara Zagora
  - Chiesi Clinical Trial - Site 100454, Stara Zagora
  - Chiesi Clinical Trial - Site 100462, Veliko Tarnovo
  - Chiesi Clinical Trial - Site 100419, Vidin
  - Chiesi Clinical Trial - Site 100457, Vidin
- Chile (6):
  - Chiesi Clinical Trial - Site 152406, Concepción
  - Chiesi Clinical Trial - Site 152407, Quillota
  - Chiesi Clinical Trial - Site 152403, Santiago
  - Chiesi Clinical Trial - Site 152404, Santiago
  - Chiesi Clinical Trial - Site 152409, Talca
  - Chiesi Clinical Trial - Site 152401, Valparaíso
- China (60):
  - Chiesi Clinical Trial - Site 156473, Baotou
  - Chiesi Clinical Trial - Site 156507, Baotou
  - Chiesi Clinical Trial - Site 156474, Beijing
  - Chiesi Clinical Trial - Site 156489, Beijing
  - Chiesi Clinical Trial - Site 156509, Beijing
  - Chiesi Clinical Trial - Site 156501, Changchun
  - Chiesi Clinical Trial - Site 156455, Changsha
  - Chiesi Clinical Trial - Site 156488, Changsha
  - Chiesi Clinical Trial - Site 156451, Chengdu
  - Chiesi Clinical Trial - Site 156490, Chengdu
  - Chiesi Clinical Trial - Site 156463, Chongqing
  - Chiesi Clinical Trial - Site 156511, Chongqing
  - Chiesi Clinical Trial - Site 156452, Guangzhou
  - Chiesi Clinical Trial - Site 156460, Guangzhou
  - Chiesi Clinical Trial - Site 156471, Guangzhou
  - Chiesi Clinical Trial - Site 156472, Guangzhou
  - Chiesi Clinical Trial - Site 156494, Guangzhou
  - Chiesi Clinical Trial - Site 156504, Guangzhou
  - Chiesi Clinical Trial - Site 156468, Haikou
  - Chiesi Clinical Trial - Site 156498, Hangzhou
  - Chiesi Clinical Trial - Site 156510, Harbin
  - Chiesi Clinical Trial - Site 156486, Hefei
  - Chiesi Clinical Trial - Site 156503, Hefei
  - Chiesi Clinical Trial - Site 156483, Hengyang
  - Chiesi Clinical Trial - Site 156512, Hohhot
  - Chiesi Clinical Trial - Site 156495, Huanghou
  - Chiesi Clinical Trial - Site 156506, Huizhou
  - Chiesi Clinical Trial - Site 156456, Jinan
  - Chiesi Clinical Trial - Site 156485, Jinhua
  - Chiesi Clinical Trial - Site 156454, Liaoyang
  - Chiesi Clinical Trial - Site 156453, Nanchang
  - Chiesi Clinical Trial - Site 156467, Nanchang
  - Chiesi Clinical Trial - Site 156484, Nanjing
  - Chiesi Clinical Trial - Site 156496, Nanjing
  - Chiesi Clinical Trial - Site 156497, Nanjing
  - Chiesi Clinical Trial - Site 156481, Pingxiang
  - Chiesi Clinical Trial - Site 156464, Qingyuan
  - Chiesi Clinical Trial - Site 156458, Shanghai
  - Chiesi Clinical Trial - Site 156461, Shanghai
  - Chiesi Clinical Trial - Site 156475, Shanghai
  - Chiesi Clinical Trial - Site 156476, Shanghai
  - Chiesi Clinical Trial - Site 156477, Shanghai
  - Chiesi Clinical Trial - Site 156487, Shanghai
  - Chiesi Clinical Trial - Site 156457, Suzhou
  - Chiesi Clinical Trial - Site 156499, Taiyuan
  - Chiesi Clinical Trial - Site 156469, Taizhou
  - Chiesi Clinical Trial - Site 156465, Tianjin
  - Chiesi Clinical Trial - Site 156480, Tianjin
  - Chiesi Clinical Trial - Site 156491, Wuhan
  - Chiesi Clinical Trial - Site 156505, Wuhan
  - Chiesi Clinical Trial - Site 156492, Wuxi
  - Chiesi Clinical Trial - Site 156493, Wuxi
  - Chiesi Clinical Trial - Site 156470, Xiangtan
  - Chiesi Clinical Trial - Site 156482, Xining
  - Chiesi Clinical Trial - Site 156478, Xinxiang
  - Chiesi Clinical Trial - Site 156466, Xuzhou
  - Chiesi Clinical Trial - Site 156479, Xuzhou
  - Chiesi Clinical Trial - Site 156508, Yanji
  - Chiesi Clinical Trial - Site 156459, Yiyang
  - Chiesi Clinical Trial - Site 156462, Zhanjiang
- Czechia (16):
  - Chiesi Clinical Trial - Site 203406, Brandýs nad Labem
  - Chiesi Clinical Trial - Site 203418, Havlíčkův Brod
  - Chiesi Clinical Trial - Site 203401, Jindřichův Hradec
  - Chiesi Clinical Trial - Site 203410, Lovosice
  - Chiesi Clinical Trial - Site 203417, Měšice
  - Chiesi Clinical Trial - Site 203404, Miroslav
  - Chiesi Clinical Trial - Site 203416, Mladá Boleslav
  - Chiesi Clinical Trial - Site 203453, Olomouc
  - Chiesi Clinical Trial - Site 203405, Prague
  - Chiesi Clinical Trial - Site 203407, Prague
  - Chiesi Clinical Trial - Site 203413, Prague
  - Chiesi Clinical Trial - Site 203415, Prague
  - Chiesi Clinical Trial - Site 203452, Prague
  - Chiesi Clinical Trial - Site 203402, Strakonice
  - Chiesi Clinical Trial - Site 203451, Tábor
  - Chiesi Clinical Trial - Site 203412, Varnsdorf
- Georgia (7):
  - Chiesi Clinical Trial - Site 268451, Tbilisi
  - Chiesi Clinical Trial - Site 268452, Tbilisi
  - Chiesi Clinical Trial - Site 268453, Tbilisi
  - Chiesi Clinical Trial - Site 268454, Tbilisi
  - Chiesi Clinical Trial - Site 268455, Tbilisi
  - Chiesi Clinical Trial - Site 268456, Tbilisi
  - Chiesi Clinical Trial - Site 268457, Tbilisi
- Germany (26):
  - Chiesi Clinical Trial - Site 276462, Bamberg
  - Chiesi Clinical Trial - Site 276405, Berlin
  - Chiesi Clinical Trial - Site 276406, Berlin
  - Chiesi Clinical Trial - Site 276410, Berlin
  - Chiesi Clinical Trial - Site 276411, Berlin
  - Chiesi Clinical Trial - Site 276415, Berlin
  - Chiesi Clinical Trial - Site 276452, Berlin
  - Chiesi Clinical Trial - Site 276453, Berlin
  - Chiesi Clinical Trial - Site 276457, Berlin
  - Chiesi Clinical Trial - Site 276456, Cottbus
  - Chiesi Clinical Trial - Site 276409, Darmstadt
  - Chiesi Clinical Trial - Site 276403, Delitzsch
  - Chiesi Clinical Trial - Site 276455, Essen
  - Chiesi Clinical Trial - Site 276404, Frankfurt
  - Chiesi Clinical Trial - Site 276401, Hamburg
  - Chiesi Clinical Trial - Site 276413, Hamburg
  - Chiesi Clinical Trial - Site 276463, Hanover
  - Chiesi Clinical Trial - Site 276417, Koblenz
  - Chiesi Clinical Trial - Site 276402, Leipzig
  - Chiesi Clinical Trial - Site 276416, Leipzig
  - Chiesi Clinical Trial - Site 276461, Leipzig
  - Chiesi Clinical Trial - Site 276407, Mainz
  - Chiesi Clinical Trial - Site 276408, Munich
  - Chiesi Clinical Trial - Site 276459, Münster
  - Chiesi Clinical Trial - Site 276418, Peine
  - Chiesi Clinical Trial - Site 276464, Schleswig
- Greece (6):
  - Chiesi Clinical Trial - Site 300406, Athens
  - Chiesi Clinical Trial - Site 300401, Heraklion
  - Chiesi Clinical Trial - Site 300403, Ioannina
  - Chiesi Clinical Trial - Site 300404, Thessaloniki
  - Chiesi Clinical Trial - Site 300405, Thessaloniki
  - Chiesi Clinical Trial - Site 300407, Volos
- Hungary (18):
  - Chiesi Clinical Trial - Site 348406, Balassagyarmat
  - Chiesi Clinical Trial - Site 348401, Budapest
  - Chiesi Clinical Trial - Site 348457, Budapest
  - Chiesi Clinical Trial - Site 348459, Budapest
  - Chiesi Clinical Trial - Site 348405, Csorna
  - Chiesi Clinical Trial - Site 348412, Edelény
  - Chiesi Clinical Trial - Site 348408, Gödöllő
  - Chiesi Clinical Trial - Site 348451, Gyula
  - Chiesi Clinical Trial - Site 348409, Monor
  - Chiesi Clinical Trial - Site 348407, Nyíregyháza
  - Chiesi Clinical Trial - Site 348413, Pécs
  - Chiesi Clinical Trial - Site 348452, Sellye
  - Chiesi Clinical Trial - Site 348458, Százhalombatta
  - Chiesi Clinical Trial - Site 348410, Szeged
  - Chiesi Clinical Trial - Site 348461, Szolnok
  - Chiesi Clinical Trial - Site 348403, Szombathely
  - Chiesi Clinical Trial - Site 348453, Tatabánya
  - Chiesi Clinical Trial - Site 348415, Törökbálint
- Israel (10):
  - Chiesi Clinical Trial - Site 376402, Ashkelon
  - Chiesi Clinical Trial - Site 376401, Beersheba
  - Chiesi Clinical Trial - Site 376408, Haifa
  - Chiesi Clinical Trial - Site 376403, Jerusalem
  - Chiesi Clinical Trial - Site 376406, Jerusalem
  - Chiesi Clinical Trial - Site 376407, Kfar Saba
  - Chiesi Clinical Trial - Site 376405, Petah Tikva
  - Chiesi Clinical Trial - Site 376404, Ramat Gan
  - Chiesi Clinical Trial - Site 376409, Tel Aviv
  - Chiesi Clinical Trial - Site 376451, Tel Litwinsky
- Italy (5):
  - Chiesi Clinical Trial - Site 380454, Brescia
  - Chiesi Clinical Trial - Site 380451, Catania
  - Chiesi Clinical Trial - Site 380453, Ferrara
  - Chiesi Clinical Trial - Site 380455, Roma
  - Chiesi Clinical Trial - Site 380452, Trieste
- Mexico (12):
  - Chiesi Clinical Trial - Site 484402, Chihuahua City
  - Chiesi Clinical Trial - Site 484410, Chihuahua City
  - Chiesi Clinical Trial - Site 484405, Córdoba
  - Chiesi Clinical Trial - Site 484452, Durango
  - Chiesi Clinical Trial - Site 484401, Guadalajara
  - Chiesi Clinical Trial - Site 484407, Guadalajara
  - Chiesi Clinical Trial - Site 484409, Guadalajara
  - Chiesi Clinical Trial - Site 484453, Guadalajara
  - Chiesi Clinical Trial - Site 484406, Mexico City
  - Chiesi Clinical Trial - Site 484403, Monterrey
  - Chiesi Clinical Trial - Site 484411, Monterrey
  - Chiesi Clinical Trial - Site 484404, Veracruz
- Netherlands (5):
  - Chiesi Clinical Trial - Site 528403, Almere Stad
  - Chiesi Clinical Trial - Site 528401, Beek
  - Chiesi Clinical Trial - Site 528404, Breda
  - Chiesi Clinical Trial - Site 528402, Heerlen
  - Chiesi Clinical Trial - Site 528405, Leeuwarden
- New Zealand (3):
  - Chiesi Clinical Trial - Site 554404, Christchurch
  - Chiesi Clinical Trial - Site 554402, Hamilton
  - Chiesi Clinical Trial - Site 554406, Wellington
- North Macedonia (8):
  - Chiesi Clinical Trial - Site 807402, Gostivar
  - Chiesi Clinical Trial - Site 807401, Prilep
  - Chiesi Clinical Trial - Site 807452, Skopje
  - Chiesi Clinical Trial - Site 807454, Skopje
  - General Hospital-Struga - Site 807405, Struga
  - General Hospital-Strumica - Site 807406, Strumica
  - Chiesi Clinical Trial - Site 807403, Tetovo
  - General Hospital - Veles - Site 807404, Veles
- Poland (24):
  - Chiesi Clinical Trial - Site 616413, Bialystok
  - Chiesi Clinical Trial - Site 616418, Bialystok
  - HolsaClinical - Gyncentrum Bielsko-Biala - Site 616460, Bielsko-Biala
  - Chiesi Clinical Trial - Site 616404, Giżycko
  - Chiesi Clinical Trial - Site 616415, Katowice
  - Chiesi Clinical Trial - Site 616422, Katowice
  - Chiesi Clinical Trial - Site 616409, Krakow
  - Chiesi Clinical Trial - Site 616411, Krakow
  - Chiesi Clinical Trial - Site 616414, Krakow
  - Chiesi Clinical Trial - Site 616455, Krakow
  - AmiCare Medical Centre - Site 616459, Lodz
  - Chiesi Clinical Trial - Site 616403, Lodz
  - Chiesi Clinical Trial - Site 616423, Lodz
  - Chiesi Clinical Trial - Site 616458, Lodz
  - Chiesi Clinical Trial - Site 616457, Lublin
  - Chiesi Clinical Trial - Site 616419, Ostrowiec
  - Chiesi Clinical Trial - Site 616456, Piaseczno
  - Chiesi Clinical Trial - Site 616406, Poznan
  - Chiesi Clinical Trial - Site 616408, Poznan
  - Chiesi Clinical Trial - Site 616401, Sosnowiec
  - Chiesi Clinical Trial - Site 616451, Tarnów
  - Chiesi Clinical Trial - Site 616402, Torun
  - Chiesi Clinical Trial - Site 616452, Wroclaw
  - Chiesi Clinical Trial - Site 616454, Wroclaw
- Romania (18):
  - Chiesi Clinical Trial - Site 642410, Bacau
  - Chiesi Clinical Trial - Site 642452, Bragadiru
  - Chiesi Clinical Trial - Site 642402, Cluj-Napoca
  - Chiesi Clinical Trial - Site 642404, Cluj-Napoca
  - Chiesi Clinical Trial - Site 642406, Cluj-Napoca
  - Chiesi Clinical Trial - Site 642408, Cluj-Napoca
  - Chiesi Clinical Trial - Site 642412, Cluj-Napoca
  - Chiesi Clinical Trial - Site 642454, Cluj-Napoca
  - Chiesi Clinical Trial - Site 642401, Constanța
  - Chiesi Clinical Trial - Site 642409, Craiova
  - Chiesi Clinical Trial - Site 642411, Craiova
  - Chiesi Clinical Trial - Site 642453, Deva
  - Chiesi Clinical Trial - Site 642414, Iași
  - Chiesi Clinical Trial - Site 642403, Oradea
  - Chiesi Clinical Trial - Site 642413, Reșca
  - Chiesi Clinical Trial - Site 642405, Timișoara
  - Chiesi Clinical Trial - Site 642407, Timișoara
  - Chiesi Clinical Trial - Site 642415, Timișoara
- Russia (35):
  - Chiesi Clinical Trial - Site 643433, Chelyabinsk
  - Chiesi Clinical Trial - Site 643417, Kazan'
  - Chiesi Clinical Trial - Site 643462, Kazan'
  - Chiesi Clinical Trial - Site 643456, Kemerovo
  - Chiesi Clinical Trial - Site 643401, Moscow
  - Chiesi Clinical Trial - Site 643413, Moscow
  - Chiesi Clinical Trial - Site 643428, Moscow
  - Chiesi Clinical Trial - Site 643460, Moscow
  - Chiesi Clinical Trial - Site 643454, Moskva
  - Chiesi Clinical Trial - Site 643416, Nizhny Novgorod
  - Chiesi Clinical Trial - Site 643403, Odintsovskiy
  - Chiesi Clinical Trial - Site 643457, Rostov-on-Don
  - Chiesi Clinical Trial - Site 643459, Rostov-on-Don
  - Chiesi Clinical Trial - Site 643404, Saint Petersburg
  - Chiesi Clinical Trial - Site 643405, Saint Petersburg
  - Chiesi Clinical Trial - Site 643406, Saint Petersburg
  - Chiesi Clinical Trial - Site 643408, Saint Petersburg
  - Chiesi Clinical Trial - Site 643410, Saint Petersburg
  - Chiesi Clinical Trial - Site 643411, Saint Petersburg
  - Chiesi Clinical Trial - Site 643412, Saint Petersburg
  - Chiesi Clinical Trial - Site 643414, Saint Petersburg
  - Chiesi Clinical Trial - Site 643419, Saint Petersburg
  - Chiesi Clinical Trial - Site 643420, Saint Petersburg
  - Chiesi Clinical Trial - Site 643423, Saint Petersburg
  - Chiesi Clinical Trial - Site 643424, Saint Petersburg
  - Chiesi Clinical Trial - Site 643431, Saint Petersburg
  - Chiesi Clinical Trial - Site 643458, Saint Petersburg
  - Chiesi Clinical Trial - Site 643451, Saint-Peterburg
  - Chiesi Clinical Trial - Site 643415, Saratov
  - Chiesi Clinical Trial - Site 643425, Saratov
  - Chiesi Clinical Trial - Site 643421, Ulyanovsk
  - Chiesi Clinical Trial - Site 643402, Voronezh
  - Chiesi Clinical Trial - Site 643407, Yaroslavl
  - Chiesi Clinical Trial - Site 643418, Yaroslavl
  - Chiesi Clinical Trial - Site 643426, Yaroslavl
- Serbia (10):
  - Kliničko Bolnički Centar Zvezdara - Site 688459, Belgrade
  - Chiesi Clinical Trial - Site 688401, Belgrade
  - Institut za Plućne Bolesti Sremska Kamenica - Site 688464, Kamenitz
  - Institute for Pulmonary Diseases of Vojvodina - Site 688466, Kamenitz
  - Klinički Centar Kragujevac - Site 688456, Kragujevac
  - Chiesi Clinical Trial - Site 688402, Kragujevac
  - Chiesi Clinical Trial - Site 688403, Kruševac
  - Chiesi Clinical Trial - Site 688404, Niš
  - Chiesi Clinical Trial - Site 688405, Niš
  - Chiesi Clinical Trial - Site 688463, Užice
- Slovakia (5):
  - Chiesi Clinical Trial - Site 703401, Bardejov
  - Chiesi Clinical Trial - Site 703452, Humenné
  - Chiesi Clinical Trial - Site 703403, Košice
  - Chiesi Clinical Trial - Site 703453, Levice
  - Chiesi Clinical Trial - Site 703402, Spišská Nová Ves
- South Africa (7):
  - Chiesi Clinical Trial - Site 710458, Benoni
  - Chiesi Clinical Trial - Site 710451, Bloemfontein
  - Chiesi Clinical Trial - Site 710456, Centurion
  - Chiesi Clinical Trial - Site 710454, Durban
  - Chiesi Clinical Trial - Site 710455, George
  - Chiesi Clinical Trial - Site 710453, Johannesburg
  - Chiesi Clinical Trial - Site 710452, Pretoria
- Spain (11):
  - Chiesi Clinical Trial - Site 724454, Barakaldo
  - Chiesi Clinical Trial - Site 724403, Barcelona
  - Chiesi Clinical Trial - Site 724457, Barcelona
  - Chiesi Clinical Trial - Site 724401, Córdoba
  - Chiesi Clinical Trial - Site 724404, Madrid
  - Chiesi Clinical Trial - Site 724405, Madrid
  - Chiesi Clinical Trial - Site 724451, Madrid
  - Chiesi Clinical Trial - Site 724455, Palma de Mallorca
  - Chiesi Clinical Trial - Site 724458, Pontevedra
  - Chiesi Clinical Trial - Site 724452, Valencia
  - Chiesi Clinical Trial - Site 724402, Zaragoza
- Turkey (Türkiye) (9):
  - Chiesi Clinical Trial - Site 792412, Adana
  - Chiesi Clinical Trial - Site 792410, Bornova
  - Chiesi Clinical Trial - Site 792415, Çanakkale
  - Chiesi Clinical Trial - Site 792408, Istanbul
  - Chiesi Clinical Trial - Site 792414, Kocaeli
  - Chiesi Clinical Trial - Site 792413, Mersin
  - Chiesi Clinical Trial - Site 792406, Pamukkale
  - Chiesi Clinical Trial - Site 792411, Yenişehir
  - Chiesi Clinical Trial - Site 792407, Zeytinburnu
- Ukraine (38):
  - LLC "Euromedservice" - Site 804463, Chernivtsi
  - Chiesi Clinical Trial - Site 804452, Chernivtsi
  - Chiesi Clinical Trial - Site 804422, Dnipro
  - Chiesi Clinical Trial - Site 804458, Dnipro
  - Ivano-Frankivsk City Clinical Hospital No. 1 - Site 804453, Ivano-Frankivsk
  - The Ivano-Frankivsk National Medical Univeristy - Site 804465, Ivano-Frankivsk
  - Chiesi Clinical Trial - Site 804402, Ivano-Frankivsk
  - Chiesi Clinical Trial - Site 804453, Ivano-Frankivsk
  - Chiesi Clinical Trial - Site 804404, Kharkiv
  - Chiesi Clinical Trial - Site 804405, Kharkiv
  - Chiesi Clinical Trial - Site 804406, Kharkiv
  - Chiesi Clinical Trial - Site 804409, Kharkiv
  - Chiesi Clinical Trial - Site 804450, Kharkiv
  - Chiesi Clinical Trial - Site 804457, Kharkiv
  - Chiesi Clinical Trial - Site 804403, Kherson
  - Chiesi Clinical Trial - Site 804421, Kiev
  - Chiesi Clinical Trial - Site 804459, Kiev
  - Municipal Non-profit Enterpirse-Regional Territorial Medical - Site 804454, Kramatorsk
  - Chiesi Clinical Trial - Site 804420, Kremenchuk
  - Chiesi Clinical Trial - Site 804451, Kryvyi Rih
  - ARENSIA Exploratory Medicine Medical Center - Site 804468, Kyiv
  - Medical Center- OkClinic of International Institute of Clinical Studies, LLC - Site 804466, Kyiv
  - Chiesi Clinical Trial - Site 804401, Kyiv
  - Chiesi Clinical Trial - Site 804408, Kyiv
  - Chiesi Clinical Trial - Site 804411, Kyiv
  - Chiesi Clinical Trial - Site 804412, Kyiv
  - Chiesi Clinical Trial - Site 804416, Kyiv
  - Chiesi Clinical Trial - Site 804460, Kyiv
  - Chiesi Clinical Trial - Site 804462, Kyiv
  - Chiesi Clinical Trial - Site 804427, Odesa
  - Limited Liability Company Medical and Diagnostic Center "Medion" - Site 804407, Poltava
  - Chiesi Clinical Trial - Site 804415, Vinnytsia
  - Chiesi Clinical Trial - Site 804417, Vinnytsia
  - Chiesi Clinical Trial - Site 804455, Vinnytsia
  - Chiesi Clinical Trial - Site 804456, Vinnytsia
  - Chiesi Clinical Trial - Site 804423, Zaporizhzhia
  - Chiesi Clinical Trial - Site 804426, Zaporizhzhya
  - Central City Hospital No.1 - Zhytomyr - Site 804467, Zhytomyr
- United Kingdom (4):
  - Chiesi Clinical Trial - Site 826410, Belfast
  - Chiesi Clinical Trial - Site 826409, Bradford
  - Chiesi Clinical Trial - Site 826411, London
  - Chiesi Clinical Trial - Site 826412, Rochdale

IPD SHARING:
Plan to Share IPD: No